CLINICAL TRIAL: NCT04654663
Title: Impact of Sarcopenia Index on Postoperative Pulmonary Complication in Elderly Patients Undergoing OPCAB: a Retrospective Study
Brief Title: Impact of Sarcopenia Index on Postoperative Pulmonary Complication in Elderly Patients Undergoing OPCAB
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1128
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Occlusive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective data collection. The aim of this study is to determine the effect of preoperative sarcopenia index on postoperative pulmonary complications in elderly patients undergoing off-pump coronary artery bypass graft surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were 65 years of age or older at the time of surgery(off-pump coronary artery bypass graft surgery)
* serum cystatin C and creatinine test results were valid within one week before surgery

Exclusion Criteria:

* Patients with chronic renal failure (estimated glomerular filtration rate less than 60)
* Patients with acute kidney injury
* Patients with respiratory tract infection within 1 month before surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients who undersent off-pump coronary artery bypass graft surgery.
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
postoperative pulmonary complications : pneumonia | During the hospitalization for surgery. This includes the entire postoperative period up to discharge, even if over 30 days.
  CXR with at least one of the following: infiltrate, consolidation, cavitation;plus at least one of the following: fever >38 °C with no other cause, white cell count <4 or>12*109 litre-1, >70 yr of age with altered mental status with no other cause;-plus at least two of the following: new purulent/ changed sputum, increased secretions/suctioning, new/worse cough/dyspnoea/tachypnoea, rales/ bronchial breath sounds, worsening gas exchange.
postoperative pulmonary complications : prolonged ventilation | During the hospitalization for surgery. This includes the entire postoperative period up to discharge, even if over 30 days.
  Indicate whether the patient had prolonged post-operative pulmonary ventilation > 24.0 hours. The hours of postoperative ventilation time include OR exit until extubation, plus any additional hours following reintubation.
postoperative pulmonary complications : reintubation | During the hospitalization for surgery. This includes the entire postoperative period up to discharge, even if over 30 days.
  Indicate whether the patient was intubated for the first time after leaving the OR from the initial procedure, or re-intubated during the hospital stay after the initial extubation.

SECONDARY OUTCOMES:
postoperative complications : Renal failure | During the hospitalization for surgery. This includes the entire postoperative period up to discharge, even if over 30 days.
  Indicate whether the patient had acute renal failure or worsening renal function resulting in ONE OR BOTH of the following:
  1. Increase in serum creatinine level 3.0 x greater than baseline, or serum creatinine level ≥4 mg/dL , Acute rise must be at least 0.5 mg/dl 2. A new requirement for dialysis postoperatively.
postoperative complications : Delirium | During the hospitalization for surgery. This includes the entire postoperative period up to discharge, even if over 30 days.
  Indicate whether the patient experienced postoperative delirium from OR Exit to ICU discharge.
postoperative complications : Reoperation due to bleeding/tamponade | During the hospitalization for surgery. This includes the entire postoperative period up to discharge, even if over 30 days.
  Indicate whether the patient was reexplored for mediastinal bleeding with or without tamponade either in the ICU or returned to the operating room.
postoperative complications : Permanent stroke | During the hospitalization for surgery. This includes the entire postoperative period up to discharge, even if over 30 days.
  Indicate whether the patient has a postoperative stroke (i.e., any confirmed neurological deficit of abrupt onset caused by a disturbance in blood supply to the brain) that was confirmed on imaging or did not resolve within 24 hours.
postoperative complications : Mortality | During the hospitalization in which the operation was performed, even if after 30 days.
  all deaths, regardless of cause, occurring during the hospitalization in which the operation was performed, even if after 30 days (including patients transferred to other acute care facilities)
postoperative complications : Mortality | After discharge from the hospital, but before the end of the 30th postoperative day.
  all deaths, regardless of cause, occurring after discharge from the hospital, but before the end of the 30th postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Lan Kwak, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided